CLINICAL TRIAL: NCT00610831
Title: Computed Radiography (CR) Data Collection for Mammography Computer Aided Detection (CAD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Issues
Sponsor: University of California, Irvine (Other)
Collaborators: Carestream Health, Inc. (Industry); Eastman Kodak Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UCI-HS-2007-5519; CH-41914 (Other Grant/Funding Number: Carestream Health)
Record Dates: First submitted 2008-01-12; First posted 2008-02-08 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DirectView CR Mammography (Experimental): Each subject will have routine clinical care imaging obtained and 4 standard mammogram views (RMLO, RCC, LMLO, LCC) using CR mammography. If routine mammograms were obtained on a day previous to enrollment in the study, those images (4 views; 2 views for mastectomy patients) will not be repeated for this study; only the CR images will be obtained.
  Interventions: Device: DIRECTVIEW CR Mammography

INTERVENTIONS:
Device: DIRECTVIEW CR Mammography — 4 views screening mammogram

SUMMARY:
The objective of this study is to collect an image library of diagnostic digital mammograms using the Carestream CR mammography system from patients who have histological-conformed breast cancer to demonstrate the clinical feasibility of this system for detection of breast cancer.

ELIGIBILITY:
Inclusion Requirements

* Women age 40 to 85
* Recommended for biopsy and BI-RADS assessment of category 4 (suspicious abnormality) or 5 (highly suggestive of malignancy)
* Able to have MLO and CC views taken
* Good general health
* Able and willing to provide a written Informed Consent

Exclusion Requirements

* Under age 40
* Pregnant or suspicious of being pregnant
* Breast implants
* Breasts too large to be adequately positioned on a 24 x 30 cassette
* Personal history of breast cancer treated with a lumpectomy
* Unable or unwilling to provide a written Informed Consent form

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To collect mammogram from patients with breast cancer using the Carestream Mammo CR device. | at completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Feig, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Breast Health Center, University of California Irvine Medical Center, Orange, California, United States